CLINICAL TRIAL: NCT03151980
Title: The Use of Sun Protection After Hamam (Turkish Bath): a Randomized, Controlled, Blinded Trial
Brief Title: The Use of Sun Protection After Hamam (Turkish Bath)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Stina Öberg, MD, PhD student, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Herlev and Gentofte Hospital
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: No Medical Condition

STUDY DESIGN:
Intervention Model Description: Each participant will be randomized to receive Hamam on either the left or the right side of the back. The other side will be left untreated. Each individual will thereafter receive a sun exposure of both the Hamam-treated skin and the untreated skin.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hamam treated skin and sun exposure (Active Comparator)
  Interventions: Procedure: Hamam treated skin and sun exposure
- Untreated skin and sun exposure (Other)
  Interventions: Other: Untreated skin and sun exposure

INTERVENTIONS:
Procedure: Hamam treated skin and sun exposure — Hamam is a skin treatment (soaping and scrubbing).
  Arms: Hamam treated skin and sun exposure
Other: Untreated skin and sun exposure — Skin that will not receive Hamam.
  Arms: Untreated skin and sun exposure

SUMMARY:
Hamam is a common spa treatment. During a Hamam, some of the outermost layer of the skin is removed. The investigators believe that partly removing a protective skin layer might increase the risk of sun burn, especially for skin that has not been exposed to sun for a long time.

The aim with this study is to assess if Hamam-treated skin is more susceptible to sun burn compared with untreated skin.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Healthy volunteers
* Skin types 1,2,3- Fitzpatrick scale
* Provided informed consent

Exclusion Criteria:

* Regular medication for a condition/disease
* Active skin disease
* Sun exposure on the back within four weeks prior to the start of the study
* History of premalignant or malignant skin lesions
* Tattoo covering more than half of the back

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-05-14 (Actual); Study Completion 2017-05-14 (Actual)

PRIMARY OUTCOMES:
Skin erythema | Baseline until 24 hours after sun exposure.
  Change in skin erythema: comparison of Hamam treated skin with untreated skin. Photographs of the skin will be assessed by computer analysis.

SECONDARY OUTCOMES:
Skin erythema | Baseline until 24 hours after sun exposure.
  Measured by a visual scale.
Pain | Baseline until 24 hours after sun exposure.
  Measured by a visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rosenberg, Professor, Study Chair — University of Copenhagen, Herlev Hospital; Stina Öberg, MD, Principal Investigator — University of Copenhagen, Herlev Hospital
Locations (1):
- Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No